CLINICAL TRIAL: NCT06282601
Title: STUDY OF THE EFFECT OF RHYTHMIC AND NON-RHYTHMIC MUSICAL PRIMING ON THE SYNTAX CAPACITY OF PRESBYACOUSTIC OLDER ADULTS
Acronym: AMORCAGE MUSIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GUIGOU - Defaye 2023
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Presbyacousie
MeSH Terms: interventions — Hearing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Presbyacusis patients (Experimental)
  Interventions: Other: Audiogram; Other: Musical priming for the syntax test; Other: Test MMSE; Other: Barcelona Music Reward Questionnaire

INTERVENTIONS:
Other: Audiogram — Tonal and vocal free-field without lip-reading
Other: Musical priming for the syntax test — Listening to music with a regular or irregular rhythm, then judging the grammaticality of 2x6 blocks of French sentences interrupted by a pause, each block presenting 4 sentences including 2 grammatically correct sentences and 2 grammatically incorrect sentences. The sentences are pronounced by a French female voice at a natural rhythm and comfortable volume.
Other: Test MMSE — test to assess a person's cognitive functions and memory capacity.
Other: Barcelona Music Reward Questionnaire — 20 questions exploring 5 main facets of the musical reward experience, with 4 items for each of the 5 facets, for which participants indicate the level of agreement using a 5-level scale, ranging from "strongly disagree" to "strongly agree".

SUMMARY:
Presbyacusis, or age-related hearing loss, is a public health problem, affecting 20% of men and 30% of women over the age of 70 according to the WHO. In the most incapacitating cases, hearing aids are required. Numerous studies have evaluated the benefits of hearing aids, particularly in terms of improved hearing and quality of life.

However, the specific effect of music on language skills has not yet been studied in hearing-impaired older adults.

In this context, it was decided to study the effect of musical priming on the syntactic abilities of adults aged 70 or older with presbyacusis.

This study is based on the hypothesis that music priming with regular music optimizes the syntax language skills of people with presbyacusis, as has already been proven in adults and normal-hearing children.

ELIGIBILITY:
Inclusion Criteria:

* No objection to participation in the study
* Men and women aged ≥ 70 years
* Patients diagnosed with presbyacusis (age-related bilateral and symmetrical sensorineural hearing loss, all stages combined), with or without the use of a bilateral hearing aid.
* If they use a hearing aid: hearing must have an average free-field fitted tonal threshold of 40 dB max and free-field fitted speech discrimination without lip-reading of 90-100% at 60dB in silence.
* MMSE score ≥ 24/30

Exclusion Criteria:

* Person under legal protection (curatorship, guardianship)
* Person under court order
* Adult unable to provide consent
* Person with a neurocognitive disorder (post-stroke, dyslexia, dyspraxia) or neuro-psychiatric disorder (dementia, autism)
* Severe sensorineural hearing loss with mean free-field threshold > 40 dB and free-field speech discrimination without lip-reading of < 90-100% at 60dB in silence
* Asymmetrical sensorineural hearing loss due to an additional cause of hearing loss on one side.

Secondary exclusion criteria:

Person with syntax disorder (discovery of sentence comprehension or production disorders during syntax test)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-08-02 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
linguistic performance test focusing on syntax. | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France